CLINICAL TRIAL: NCT07103460
Title: The Effect of Essential Oil Diffusion Combined With Respiratory Training on the Respiratory Function of Patients With Acute Pulmonary Infections and Type 2 Diabetes
Brief Title: Essential Oil-Assisted Respiratory Training in Type 2 Diabetic Patients With Lung Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Yu-Shan Hsieh, Associate professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: B2023051651
Record Dates: First submitted 2025-07-19; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Pulmonary Infections; Pneumonia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Combination Product: Essential Oil Diffusion Combined with Respiratory Training

INTERVENTIONS:
Combination Product: Essential Oil Diffusion Combined with Respiratory Training — three commonly used essential oils (wintergreen, peppermint, and eucalyptus) will be integrated into IS respiratory training

SUMMARY:
Previous studies have shown that baseline pulmonary function in patients with type 2 diabetes mellitus (T2DM) is approximately 8% to 10% lower than in healthy individuals. Under similar infection conditions, respiratory function impairment is more pronounced in T2DM patients. Therefore, this project aims to explore the effects of incentive spirometry (IS) respiratory training combined with an essential oil diffusion device on improving respiratory function in T2DM patients. Over next two years, this study will utilize data from medical history, blood examination, cardiopulmonary endurance evaluations, subjective respiratory symptom assessments, and pulmonary function analyses to demonstrate the improving effect of the intervention in the patients with T2DM and pulmonary infection. In the first year, the study will focus on assessing the improvement in respiratory function among T2DM patients with concurrent pulmonary infections following IS respiratory training. In the second year, three commonly used essential oils (wintergreen, peppermint, and eucalyptus) will be integrated into IS respiratory training. The goal is to enhance patient comfort during training while improving the effectiveness of respiratory training and investigating the mechanisms and effects of different essential oils. The expected outcomes of this study include demonstrating that IS respiratory training combined with an essential oil diffusion device developed by our research team, could more effectively improve the respiratory function of T2DM patients with pulmonary infections. Building on this foundation, the project aims to increase patient comfort during training sessions by incorporating three commonly available essential oils-wintergreen, peppermint, and eucalyptus. This approach is expected to enhance patient acceptance of respiratory training interventions, laying a solid foundation for clinical promotion. Additionally, the study will analyze the differential effects of these essential oils on respiratory function improvement, providing a cornerstone for future clinical research in the fields of chemistry,

ELIGIBILITY:
Inclusion Criteria:

I. Currently hospitalized due to pulmonary infection (ICD-10 codes: J00.x to J22.x).

II. Diagnosed with type 2 diabetes mellitus (ICD-10 codes: E10.x or E11.x). III. Aged between 18 and 90 years. IV. Able to communicate verbally or non-verbally and understand Mandarin or Taiwanese.

V. Willing to participate in the study and consent to group assignment.

Exclusion Criteria:

I. Modified Rankin Scale (mRS) score ≥ 5, indicating severe functional impairment.

II. Diagnosed with dementia (unable to comprehend or follow intervention instructions).

III. Presence of acute psychiatric symptoms that impair communication. IV. Individuals with high litigation risk. V. Diagnosed with chronic obstructive pulmonary disease (COPD) or any other chronic respiratory diseases.

VI. Diagnosed with glucose-6-phosphate dehydrogenase (G6PD) deficiency (ICD-10 codes: D55.x, D74-75.x).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
fasting sugar (mg/dl) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  A fasting blood sugar test measures the amount of glucose in blood after you haven't eaten for at least 8 hours. The test is typically performed first thing in the morning before breakfast.
Glycated Hemoglobin; HbA1c (%) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  Glycated hemoglobin, also known as HbA1c, is a blood test that reflects average blood sugar levels over the past 2-3 months. It measures the percentage (%) of red blood cells coated with glucose (sugar).
Oxyhemoglobin saturation by pulse oximetry; SpO2 (%) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  SpO2, or peripheral oxygen saturation, is the percentage of hemoglobin in blood that is carrying oxygen, as measured by a pulse oximeter. It's a non-invasive way to estimate how much oxygen is in blood, with normal levels typically ranging from 95-100%.
Hemoglobin; Hb(g/dL) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  Hemoglobin (Hb) is a protein found in red blood cells that carries oxygen throughout the body. The amount of hemoglobin in the blood is measured and expressed in grams per deciliter (g/dL).
lactate(mmol/L) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  Lactate, also known as lactic acid, is a molecule produced during the breakdown of glucose for energy, particularly when oxygen is limited.
  The common unit for lactate is millimoles per liter (mmol/L). In clinical tests, lactate concentration is usually expressed in this unit.
Dyspnea-12 score; D-12 | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  D-12-C scale was developed, which demonstrated satisfactory reliability and validity in measuring dyspnoea among COPD patients.D-12 consists of 12 descriptor items on a scale of none (0), mild (1), moderate (2), or severe (3). Higher scores indicate more severe dyspnea.
Pulmonary function test-PEF (peak expiratory flow)(L/min) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  Peak expiratory flow (PEF) or peak expiratory flow rate (PEFR) measures how quickly you can blow air out of your lungs. It's a way to assess how well your lungs are working, particularly for those with asthma or other lung conditions. A peak flow meter, a handheld device, is used to measure it.
lung function test- FEV1(Forced expiratory volume in the first second ) (L) | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  FEV1, or Forced Expiratory Volume in 1 second, is a measurement used in lung function tests, specifically spirometry. It represents the amount of air a person can forcefully exhale in the first second of a forced exhalation after taking a deep breath. The unit for FEV1 is liters (L)

OTHER OUTCOMES:
Six-Minute walk test; 6MWT | baseline(admission), pre-intervention (1-24hrs, before intervention) and post-intervention (1-24hrs, after intervention)
  The 6-minute walk test (6MWT) is a simple, submaximal exercise test used to assess a patient's functional exercise capacity. It measures how far a person can walk in six minutes on a flat, hard surface (meter).

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital Songshan Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided